CLINICAL TRIAL: NCT06487676
Title: Long Term Follow up of Toe-to-hand Transfers: Validated Patient Reported Outcomes
Brief Title: Long Term Follow up of Toe-to-hand Transfers
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505775B0C104
Record Dates: First submitted 2024-05-05; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-05

CONDITIONS: Toe Transfer; Free Tissue Flap; Patient Reported Outcome Measures
MeSH Terms: interventions — Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Toe transfer: Patients who have undergone toe to hand transfer
  Interventions: Procedure: Toe transfer
- Replantation: Patients who have undergone finger replantation
  Interventions: Procedure: Replantation

INTERVENTIONS:
Procedure: Toe transfer — Toe-to-hand transfer
  Groups: Toe transfer
Procedure: Replantation — Finger or thumb replantation after amputation
  Other Names: Finger or thumb replantation
  Groups: Replantation

SUMMARY:
Toe transfers are perceived to have changed the landscape of the injured hand over the last half century, yet there are limited validated data that unequivocally support the functional role of toe transfers after traumatic digital amputation. There also remain unanswered questions about what factors critically influence functional outcomes, be it sensory recovery, grip strength or other modality. Furthermore, the use of validated patient reported outcome measures (PROMs) in large series of toe transfers with long term follow up, is lacking.

DETAILED DESCRIPTION:
Finger amputations are associated with profound impacts on physical, socio-economic, vocational and mental well-being. Thumb amputations account for the greatest burden of disability globally amongst hand trauma.

The multi-centre FRANCHISE study and a recent large prospective multi-centre study have demonstrated that finger replantation outperforms equivalent amputations in nearly all digits at all levels, except for the little finger. However, one crucial question in hand surgery is whether toe transfers can provide a similar functional benefit to replantation.

Finger amputations are frequently not replantable even with timely access to specialized reconstructive care. A review of replantation in the USA found that of 3,417 digital amputations, only 631 replantations were attempted (18%), and of these 30% failed. Therefore nearly 90% of patients with finger amputations will ultimately live without the amputated digit.

Microvascular toe-to-hand transfer, first described in the 1960s, has a success rate close to 100% in high volume centres. There are few validated data that support the functional benefits of toe transfer, with the majority of outcome studies focusing on operative survival rates, physical measurements such as grip strength, or employ unvalidated scales and self-created questionnaires. More data, in larger more representative populations, using validated PROMs, is required.

Here, we aim to demonstrate using PROMS that the role of toe transfers has equivalent or improved functional benefits, with comparison to finger replantation. Additionally, this study aims to identify physical factors that have the greatest influence on patient reported outcomes. This may answer fundamental questions regarding optimum strategies for the design of toe transfers.

ELIGIBILITY:
Inclusion Criteria:

* Toe transfers
* minimum 5 year follow up

Exclusion Criteria:

* partial toe transfers including toenail, toe pulp or vascularised joint
* under 5 year follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated on by single surgeon (FCW) at Chang Gung Memorial Hospital from 1983 to 2015, with at least 5 years follow up at time of inclusion to study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Michigan Hand Questionnaire | Single time-point, on average 22 years after surgery
  Validated Hand function patient reported outcome measured. 0-100. Higher is better

SECONDARY OUTCOMES:
Short Form 36 | Single time-point, on average 22 years after surgery
  Short Form 36 Quality of Life. 0-100. Higher is better
Foot Function Index | Single time-point, on average 22 years after surgery
  Validated foot function Patient reported outcome measure. 0-100. Lower is better
Aesthetic evaluation | Longitudinal. 3 timepoints: 1 day before surgery, 1 day after surgery, and on average 22 years after surgery
  Subjective evaluation of toe transfer appearance using a Visual Analogue Scale, not validated

OTHER OUTCOMES:
Range of motion | Single time-point, on average 22 years after surgery
  Total active range of motion of digit. Measured in degrees per digit
Grip strength | Single time-point, on average 22 years after surgery
  Measured with hand dynamometer. Measured in kilograms.
Sensation | Single time-point, on average 22 years after surgery
  Measured with discriminator device. Two point discrimination measured in millimetres

CONTACTS AND LOCATIONS:
Overall Officials: Fu Chan Wei, FACS, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Data subject to privacy and legal restrictions - not yet decided